CLINICAL TRIAL: NCT05728632
Title: Cardioprotective Effects of Nebivolol Versus Placebo in Patients Undergoing Chemotherapy With Anthracyclines (CONTROL Trial)
Brief Title: Cardioprotective Effects of Nebivolol Versus Placebo in Patients Undergoing Chemotherapy With Anthracyclines
Acronym: CONTROL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Giulio Stefanini (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor-Investigator, Giulio Stefanini, Professor, Humanitas Hospital, Italy
Organization: Humanitas Hospital, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 012018CONTROL
Record Dates: First submitted 2023-01-25; First posted 2023-02-15 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Lymphoma, Large B-Cell, Diffuse; Cardiotoxicity; Left Ventricular Dysfunction; Chemotherapy Effect
Keywords: anthracycline chemotherapy; nebivolol; cardio-oncology; cancer therapy-related cardiovascular toxicity; cardiac magnetic resonance; primary prevention; cardioprotection; cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Lymphoma, Large B-Cell, Diffuse; Cardiotoxicity; Ventricular Dysfunction, Left | interventions — Nebivolol

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, treating physicians, investigators, and outcome assessors are masked to the allocated treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebivolol (Experimental): nebivolol, capsule, 5 mg once daily, for 12 months
  Interventions: Drug: Nebivolol
- Placebo (Placebo Comparator): placebo, capsule, once daily, for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol — Nebivolol, capsule, 5 mg once daily, for 12 months
  Other Names: Lobivon
  Arms: Nebivolol
Drug: Placebo — Placebo, capsule, once daily, for 12 months
  Arms: Placebo

SUMMARY:
As the cancer-related prognosis improves thanks to recent advances in cancer-targeted therapies, the prognostic burden of chemotherapy-related complications - including cardiotoxicity - is increasingly recognised. So far, the evidence supporting pharmacological preventive strategies in cardio-oncology has been inconsistent and conflicting, and there is a clear need for well-designed trials with novel interventions. In this study, by using cardiac magnetic resonance, the investigators want to assess if a commonly used beta-blocker with a unique pharmacological profile, i.e. nebivolol, can prevent cardiac dysfunction in patients with breast cancer or diffuse large B-cell lymphoma undergoing chemotherapy with anthracyclines.

DETAILED DESCRIPTION:
During the last decades, major efforts have been made in the field of cancer therapy to improve prognosis and quality of life of patients treated with any sort of chemotherapy. Cardiotoxicity represents one of the most relevant adverse effects of chemotherapy, primarily in patients treated with anthracyclines. The potential protective role of cardiovascular medications in the prevention of cardiotoxicity associated with anthracyclines chemotherapy is still a matter of debate since evidence in this field are scarce and largely inconclusive. Indeed, prior studies were often limited by a non-blinded design or an echocardiography-based assessment of left ventricular ejection fraction (with a relevant inter and intra-operator variability). The primary objective of the trial is to evaluate the cardioprotective effects of the betablocker nebivolol in an individually randomized, parallel, placebo-controlled, double-blinded (patient, treating physician, investigator, outcomes assessor, statistician), superiority trial in patients with a solid tumor (i.e., breast cancer) or a hematologic malignancy (i.e., diffuse large B cell lymphoma) who have a normal cardiac function as assessed by echocardiography and will receive anthracyclines as part of their first-line chemotherapy program. Indeed, recent evidence suggests that anthracycline cardiotoxicity seems mainly due to an anthracycline-induced dysregulation of mitochondrial activity and metabolism in cardiomyocytes. Nebivolol has a distinctive profile among beta-blockers, with the unique power of increasing the nitric oxide bioavailability. Nebivolol-induced nitric oxide release has shown favourable effects in terms of antioxidant activity, cardiac neo-angiogenesis, mitochondrial and endothelial protection. On this basis, the individually randomized, parallel, placebo-controlled, double-blinded (patient, treating physician, investigator, outcomes assessor, statistician), superiority CONTROL trial will assess the cardioprotective effects of a commonly used betablocker (nebivolol) in patients with baseline normal left ventricular systolic function receiving anthracycline chemotherapy as first-line chemotherapy for breast cancer or diffuse large B-cell lymphoma. The assessment of left ventricular ejection fraction and related endpoints will be performed with cardiac magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Established histologic diagnosis of breast cancer or diffuse large B-cell lymphoma
* Planned chemotherapy with anthracyclines
* left ventricular ejection fraction ≥55% (assessed by echocardiography)
* Ability to provide informed consent

Exclusion Criteria:

* Known intolerance/contraindications to betablocker therapy
* History of coronary artery disease
* History of cardiomyopathy
* History of heart failure
* Ongoing treatment with betablockers for other indications
* Heart rate at baseline <60 beats per minute
* Arterial blood pressure at baseline <100/60 mmHg
* Contraindications to undergo cardiac magnetic resonance (e.g., non-compatible pacemakers or metallic prosthesis)
* Pregnancy or lactation
* Current participation to another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction reduction assessed by Cardiac Magnetic Resonance | from baseline to 12 months
  The primary endpoint is defined as Left Ventricular Ejection Fraction (LVEF) reduction (unit of measurement: %) assessed by Cardiac Magnetic Resonance at 12 months of follow-up.
  LVEF reduction is defined as the difference between LVEF at baseline and LVEF at 12 months follow-up (LVEF reduction = Baseline LVEF - 12 months LVEF).

SECONDARY OUTCOMES:
Left ventricular ejection fraction assessed by Cardiac Magnetic Resonance | at 12-month follow-up
  Left ventricular ejection fraction (unit of measurement: %) assessed by Cardiac Magnetic Resonance at 12-month follow-up.
Myocardial fibrosis assessed by Cardiac Magnetic Resonance | at 12-month follow-up
  Myocardial fibrosis assessed by Cardiac Magnetic Resonance with T1-mapping sequences and with Late Gadolinium Enhancement images.
Myocardial edema assessed by Cardiac Magnetic Resonance | at 12-month follow-up
  Myocardial edema assessed by Cardiac Magnetic Resonance with T2 sequences.
Right ventricular ejection fraction assessed by Cardiac Magnetic Resonance | at 12-month follow-up
  Right ventricular ejection fraction (unit of measurement: %) assessed by Cardiac Magnetic Resonance
Left ventricular end-diastolic volume assessed by Cardiac Magnetic Resonance | at different timepoints (1-month, 6-month, 12-months)
  Left ventricular end-diastolic volume (unit of measurement: ml) assessed by Cardiac Magnetic Resonance
Left ventricular end-systolic volume assessed by Cardiac Magnetic Resonance | at different timepoints (1-month, 6-month, 12-months)
  Left ventricular end-systolic volume (unit of measurement: ml) assessed by Cardiac Magnetic Resonance
Left ventricular mass assessed by Cardiac Magnetic Resonance | at different timepoints (1-month, 6-month, 12-months)
  Left ventricular mass (unit of measurement: g/m²) assessed by Cardiac Magnetic Resonance
Left ventricular ejection fraction assessed by Echocardiography | at different timepoints (1-month, 6-month, 12-months)
  Left ventricular ejection fraction (unit of measurement: %) assessed by Echocardiography
Left ventricular diastolic function assessed by Echocardiography | at different timepoints (1-month, 6-month, 12-months)
  Left ventricular diastolic function assessed by Echocardiography according to Guidelines of European Association of Cardiovascular Imaging / American Society of Echocardiography
Right ventricular systolic function assessed by Echocardiography | at different timepoints (1-month, 6-month, 12-months)
  Right ventricular systolic function assessed by Echocardiography according to Guidelines of European Association of Cardiovascular Imaging / American Society of Echocardiography
Left ventricular end-diastolic volume assessed by Echocardiography | at different timepoints (1-month, 6-month, 12-months)
  Left ventricular end-diastolic volume (unit of measurement: ml) assessed by Echocardiography
Left ventricular end-systolic volume assessed by Echocardiography | at different timepoints (1-month, 6-month, 12-months)
  Left ventricular end-systolic volume (unit of measurement: ml) assessed by Echocardiography
Serum troponin | at different timepoints (1-month, 6-month, 12-months)
  Serum high-sensitivity cardiac troponin I levels (unit of measurement: ng/L)
Serum B-type natriuretic peptide (BNP) | at different timepoints (1-month, 6-month, 12-months)
  Serum B-type natriuretic peptide (BNP) (unit of measurement: pg/mL)
Serum N-terminal-pro hormone B-type natriuretic peptide (NT-proBNP) | at different timepoints (1-month, 6-month, 12-months)
  Serum N-terminal-pro hormone B-type natriuretic peptide (NT-proBNP) levels (unit of measurement: pg/mL)
All-cause mortality | at 12-month follow-up
  All-cause mortality
Cardiovascular mortality | at 12-month follow-up
  Cardiovascular mortality or death will be defined as any death due to immediate cardiovascular cause (e.g. myocardial infarction, low-output failure, arrhythmia). Unwitnessed death and death of unknown cause will be classified as cardiac death.
Myocardial infarction | at 12-month follow-up
  Myocardial infarction will be defined according to the 3rd Universal Definition.
Cerebrovascular events | at 12-month follow-up
  Cerebrovascular events will be defined as follows:
  * Transient ischemic attack: rapidly developed clinical signs of global disturbance of cerebral function lasting fewer <24 hours, regardless of the presence of an acute clinically relevant brain lesion in imaging.
  * Ischemic stroke: rapidly developed clinical signs of focal or global disturbance of cerebral function lasting >24 hours with imaging of an acute clinically relevant brain lesion.
  * Intracerebral haemorrhage: diagnosis must be confirmed by cerebral imaging.
Hospitalization for heart failure | at 12-month follow-up
  Hospitalization for heart failure will be defined as any unplanned hospital readmission due to signs and symptoms of heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Condorelli, MD,PhD,Prof, Principal Investigator — IRCCS Humanitas Research Hospital, Rozzano-Milan, Italy; Giulio G Stefanini, MD,PhD,Prof, Principal Investigator — IRCCS Humanitas Research Hospital, Rozzano-Milan, Italy; Carmelo Carlo-Stella, MD,Prof, Principal Investigator — IRCCS Humanitas Research Hospital, Rozzano-Milan, Italy
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, Milan, Italy

REFERENCES:
- [Derived] Cannata F, Stefanini G, Carlo-Stella C, Chiarito M, Figliozzi S, Novelli L, Lisi C, Bombace S, Panico C, Cosco F, Corrado F, Masci G, Mazza R, Ricci F, Monti L, Ferrante G, Santoro A, Francone M, da Costa BR, Juni P, Condorelli G. Nebivolol versus placebo in patients undergoing anthracyclines (CONTROL Trial): rationale and study design. J Cardiovasc Med (Hagerstown). 2023 Jul 1;24(7):469-474. doi: 10.2459/JCM.0000000000001491. PMID 37285278